CLINICAL TRIAL: NCT04586777
Title: Effects of Transvertebral Direct Current Stimulation in Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Relocation of PI
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 44067
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries; Paraplegia and Tetraplegia
Keywords: neuroplasticity; transvertebral direct current stimulation; transspinal direct current stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tvDCS (Experimental): 20 minutes of anodal tvDCS will be applied over the spine at 2.5mA.
  Interventions: Device: transvertebral direct current stimulation (tvDCS)
- Cathodal tvDCS (Experimental): 20 minutes of cathodal tvDCS will be applied over the spine at 2.5mA.
  Interventions: Device: transvertebral direct current stimulation (tvDCS)
- Sham tvDCS (Sham Comparator): 20 minutes of sham tvDCS will be applied over the spine.
  Interventions: Device: transvertebral direct current stimulation (tvDCS)

INTERVENTIONS:
Device: transvertebral direct current stimulation (tvDCS) — tvDCS is a painless, non-invasive form of spinal stimulation which delivers safe, low levels of electrical current to the spinal cord through the back. It is believed to be able to influence the excitability of the brain and spinal cord.

SUMMARY:
This study will evaluate the effects of non-invasive stimulation of the spinal cord in people with spinal cord injury.

DETAILED DESCRIPTION:
This study will use a non-invasive form of spinal stimulation, called transvertebral direct current stimulation, or tvDCS. It currently is not clear what effects this type of stimulation has on the excitability of the brain and spinal cord in people with spinal cord injury. In this study, subjects will participate in 3 sessions, with at least 1 week in between sessions, during which they will get a different condition of tvDCS. We will test the excitability of the brain and spinal cord before and after tvDCS in each session.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Motor incomplete spinal cord injury classified as B, C, or D by the American Spinal Injury Association Impairment Scale (AIS)
* More than 12 months post-injury
* Lesion at of above thoracic level T8
* Body mass index <30 (in order to facilitate reliable location of body landmarks guiding stimulation)
* Severe gait deficit

Exclusion Criteria:

* Unstable cardiopulmonary conditions
* History of seizure, head injury with loss of consciousness, severe alcohol or drug abuse, and/or psychiatric illness
* Cognitive deficits severe enough to preclude informed consent
* Positive pregnancy test of being of childbearing age and not using appropriate contraception
* Ferromagnetic material in the brain or in the spine (except for titanium for segmental fixation of the spine)
* Cardiac or neural pacemakers
* Fixed contractures in the lower extremities
* Uncontrolled diabetes
* Severe osteoporosis
* Severe spasticity
* Decubitus ulcers which interfere with harness support or walking
* Severe orthostatic hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Change in corticospinal excitability | Immediately before tvDCS, Immediately after tvDCS
  This will be measured using transcranial magnetic stimulation to evoke responses in muscles of the lower leg.
Change in spinal cord excitability | Immediately before tvDCS, Immediately after tvDCS
  Hoffmann's reflex will be used to assess spinal cord excitability. For this text, pulses of electrical stimulation will be applied to the back of the knee and the response will be measured from the calf muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky at Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No